CLINICAL TRIAL: NCT02487732
Title: Comparison of Ticagrelor vs. Prasugrel on Inflammation, Arterial Stiffness, Endothelial Function, and Circulating Endothelial Progenitor Cells in Diabetic Patients With Non-ST Elevation Acute Coronary Syndrome (NSTE-ACS) Requiring Coronary Stenting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Soon Jun Hong, Associate Professor, Korea University Anam Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Adenosine diphosphate blockers
Record Dates: First submitted 2015-06-27; First posted 2015-07-01 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Acute Coronary Syndrome
Keywords: Diabetic Patients With Non-ST Elevation
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Ticagrelor; Prasugrel Hydrochloride

ARMS (2):
- Ticagrelor (Active Comparator): 180mg loading dose, 90mg twice daily for 5 weeks, then crossover to prasugrel
  Interventions: Drug: Ticagrelor
- Prasugrel (Active Comparator): 60mg loading dose, 10mg once daily for 5 weeks, then crossover to ticagrelor
  Interventions: Drug: Prasugrel

INTERVENTIONS:
Drug: Ticagrelor — Ticagrelor 90mg twice daily for 5 weeks
  Other Names: Brilinta
  Arms: Ticagrelor
Drug: Prasugrel — Prasugrel 10mg once daily for 5 weeks
  Other Names: Effient
  Arms: Prasugrel

SUMMARY:
To investigate pleiotropic effects of ticagrelor in addition to its antiplatelet effects in type 2 diabetic patients with non-ST elevation acute coronary syndrome by measuring inflammatory markers, circulating number of endothelial progenitor cells, brachial artery endothelial function, and arterial stiffness.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Newly diagnosed type 2 diabetic patients or type 2 diabetic patients on hypoglycemic agents between the age of 30 to 70
3. Non-ST elevation Acute coronary syndrome with successful coronary stent implantation (with TIMI flow grade 3 after the procedure)

Exclusion Criteria:

1. Hypersensitivity to ticagrelor, prasugrel or any of the excipients
2. No prior use of either ticagrelor or prasugrel within a month prior to randomization.
3. History of intracranial bleeding at any time
4. Active pathologic bleeding
5. Hemoglobin A1c >9%
6. Type 1 diabetes
7. Decreased serum platelet level (< 100,000/uL)
8. Need for chronic oral anticoagulant therapy or chronic low-molecular-weight heparin
9. Gastrointestinal bleed within the past 6 months, or major surgery within 30 days
10. Renal failure requiring dialysis or anticipated need for dialysis during the course of the study
11. Any condition which in the opinion of the investigator would make it unsafe or unsuitable for the patient to participate in this study
12. Involvement in the planning and/or conduct of the study
13. Left ventricular ejection fraction < 40%
14. Hepatic dysfunction (aspartate aminotransferase or alanine aminotransferase > twice the upper limit)
15. Gastrointestinal disorder such as Crohn's disease
16. Alcohol abuse
17. Steroid or hormone replacement therapy
18. Serum creatinine > 2.0 mg/dL.
19. Prior history of CVA or stroke
20. Body weight < 60 kg
21. Life expectancy less than a year
22. Known pregnancy, breast-feeding, or intend to become pregnant during the study period

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-07; Primary Completion 2016-08 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Changes in circulating number of endothelial progenitor cells | Expected average of 5 weeks
Changes in brachial artery flow mediated dilation | Expected average of 5 weeks

SECONDARY OUTCOMES:
Composite measure of brachial-ankle pulse wave velocity, and augmentation index. | Expected average of 5 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Jeong HS, Hong SJ, Cho SA, Kim JH, Cho JY, Lee SH, Joo HJ, Park JH, Yu CW, Lim DS. Comparison of Ticagrelor Versus Prasugrel for Inflammation, Vascular Function, and Circulating Endothelial Progenitor Cells in Diabetic Patients With Non-ST-Segment Elevation Acute Coronary Syndrome Requiring Coronary Stenting: A Prospective, Randomized, Crossover Trial. JACC Cardiovasc Interv. 2017 Aug 28;10(16):1646-1658. doi: 10.1016/j.jcin.2017.05.064. PMID 28838475